CLINICAL TRIAL: NCT05152719
Title: Effect of Sprint Interval Training and Intermittent Fasting on Cognitive Function
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Western University, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 119418
Record Dates: First submitted 2021-10-03; First posted 2021-12-10 (Actual); Last update posted 2021-12-10 (Actual); Status verified 2021-06

CONDITIONS: Cognitive Function

STUDY DESIGN:
Intervention Model Description: This study will include participants aged 18-39, 3 conditions analyzed for cognitive function and body composition. It will involve 120 participants randomly assigned to one of three groups with either sprint interval training, time restricted eating, or both. The study will be 6 weeks in duration.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sprint Interval Training (SIT) Protocol (Experimental): Participants in the SIT group will start with a 5 minute warm-up jogging at around 70-80% of their heart rate max. The SIT protocol consists of 30 second intervals of "all out" shuttle runs, seperated by 2 minutes of low pace walking active rest. This will be repeated between 4 times during the first 2 weeks, 5 times during the second 2 weeks, and 6 times during the third 2 weeks. Participants will be instructed to sprint the greatest possible distance in 30 seconds, starting by running to the 5m marker and back, then to the 10m marker and back, then to the 15m marker etc. The SIT session will finish with 2 minutes walking at a pace 50% of their heart rate max.
  Interventions: Behavioral: Cognitive Performance
- Time Restricted Eating (TRE) Protocol (Active Comparator): Participants will be asked to limit their food intake to the hours between 12pm to 8pm, and fast outside of these hours. During the fast, participants may consume zero calorie beverages with no caffeine or artificial sweetener. Participants are instructed to maintain their diet, with no restrictions on the type or amount of food consumed in the feeding window.
  Interventions: Behavioral: Cognitive Performance
- Combined Sprint Interval Training (SIT) and Time Restricted Eating (TRE) Protocol (Active Comparator): Participants will be asked to abide by the same eating regimen as the Time Restricted Eating Protocol Arm. Additionally, participants in this arm will perform the SIT protocol, in the fasted state. The SIT protocol will be identical to that listed in the Sprint Interval Training Protocol Arm.
  Interventions: Behavioral: Cognitive Performance

INTERVENTIONS:
Behavioral: Cognitive Performance — Cognitive function will be measured biweekly 20 minutes after exercise, or at a matched time for the Time Restricted Eating Protocol arm. The Stroop test will be completed on Mondays and the Corsi block test will be completed on Wednesdays. Body composition will be measured on Fridays using a BodPod at baseline, week 3, and week 6.

SUMMARY:
Several lifestyle modifications, such as manipulating diet and exercise, have been shown to enhance cognitive function. This study aims to determine if a combination of Sprint Interval Training (SIT) and Time Restricted Eating (TRE) elicits greater enhancements in cognitive function than either of these interventions alone. SIT and TRE have both been proven to have high adherence rates and require minimal lifestyle changes, therefore the implementation of these may allow for a feasible method of improving cognition in healthy populations. A group of young adults will be randomized into either a SIT group, TRE group, or a SIT+TRE group. To assess the changes in cognitive function, cognitive tests will be performed at baseline and biweekly. Secondly, we will be monitoring the differences in the three groups in terms of body composition, which will be measured using a BodPod. It is hypothesized that the SIT+TRE group will display the greatest improvements in cognitive function and body composition versus the TRE only group and the SIT only group.

DETAILED DESCRIPTION:
This study will explore how a combination of a time restricted eating (TRE) strategy and a sprint interval training (SIT) exercise program will affect cognitive function. Both TRE and SIT have been shown to present significant brain challenges, and are both easily implemented lifestyle habits. Participants will be randomized into 3 groups of either SIT alone, TRE alone, or SIT + TRE. We will be assessing acute effects (single day of TRE, followed by a single session of SIT the next day), and the effects over a 6 week period. The SIT protocol consists of four 30 second sprinting bouts, separated by 2 minutes of recovery. An additional sprint bout will be added biweekly to maintain progressive overload. SIT will be performed 3 times a week for the treatment group. The TRE involves no restrictions on the type or amount of food consumed, however, food must be consumed between 12pm and 8pm. The SIT will occur in an unfed state towards the end of the fast. The study will involve sedentary young adults. To evaluate the success of the intervention, 2 cognitive tests (Stroop and Corsi block) will be performed at baseline and biweekly over a 6 week treatment period. Additionally, body composition testing will occur at baseline and once every three weeks using a BodPod. We hypothesize that the combination treatment group will have greater improvements in their cognitive function and body composition compared to either intervention alone.

ELIGIBILITY:
Inclusion Criteria:

* Between 18-39 years old
* Sedentary (not meeting 50 minutes of moderate to vigorous physical activity per week)
* Pass the Physical Activity Readiness (PARQ) questionnaire

Exclusion Criteria:

* Have diabetes (self-reported)
* Have a history of smoking (self-reported)
* Take medication for weight loss (self-reported)
* Are pregnant, become pregnant, or are breastfeeding during the study (self-reported)
* Physical activity >50 minutes of moderate to vigorous physical activity per week
* Unstable weight during the 6 months prior to commencement of study (>4kg weight loss/gain)
* Have uncontrolled hypertension blood pressure >160/90
* Have a history of heart disease, previous myocardial infarction, or stroke
* Have participated in a sprint interval training exercise program in the past 6 months
* Have participated in regular intermittent fasting (≥2 weeks) in the past 6 months
* Have BMI under 18.5 or over 30

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-12-02 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Stroop Performance | 6 Weeks
  Participants' performance on the Stroop test

SECONDARY OUTCOMES:
Corsi Block Performance | 6 Weeks
  Participants' performance on the Corsi block test

OTHER OUTCOMES:
Body Composition | 6 Weeks
  Participants' body fat percentage as measured using a BodPod

CONTACTS AND LOCATIONS:
Locations (1):
- Exercise Nutrition Laboratory (Western University), London, Ontario, Canada